CLINICAL TRIAL: NCT07116135
Title: Speech Understanding and Listening Effort Benefits of Infinio Sphere
Brief Title: Speech Understanding and Listening Effort Benefits of Hearing Instruments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-22934 STUDY7873
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-01

CONDITIONS: Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Bilateral | interventions — Hearing Aids

STUDY DESIGN:
Masking Description: The participant will not know which condition they are being tested in, but all participants will be given the same intervention and not blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hearing instrument users (Experimental): Individuals with hearing impairment will be fit with three different models of hearing instruments. They will all be fit with the same hearing instruments, although they will not be aware which model they are using at the time of testing.
  Interventions: Device: hearing instruments

INTERVENTIONS:
Device: hearing instruments — Participants will be fit with three different models of hearing instruments.
  Other Names: hearing aids

SUMMARY:
The goal of this clinical study is to investigate the benefits of hearing instrument use in adults with hearing loss. The main questions it aims to answer are:

Does hearing instrument use improve speech understanding and listening effort amount people with hearing loss? Researchers will compare varying models of hearing instruments to see how speech understanding and listening effort are impacted.

Participants will be asked to wearing varying hearing instruments and participate in lab-based activities to evaluate their speech understanding, listening effort, and subjective preference.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-95 years
* N3 or N4 hearing loss
* Experienced hearing aid user
* English fluency
* Cognitively able to complete complex listening tasks

Exclusion Criteria:

* Outside of specified age range
* Vulnerable populations
* Hearing within normal limits or otherwise not appropriate for hearing instruments under study
* Inability to read, write, or speak English
* Inability to complete complex listening tasks

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Speech intelligibility as assessed by the Coordinate Response Measure (CRM) Task | Data is collected during the second lab visit for each participant, approximately 2 weeks after study enrollment. The duration of the study visit including testing is approximately 2.5 hours.
  During the CRM task (Bolia et al., 2000), participants are presented with a phrase detailing the following identifiers: target, color, and digit.
  They must listen for a target name and respond with the corresponding color and digit. Speech intelligibility performance is assessed based on accuracy, or percent correct across all trials conducted in a given condition.

SECONDARY OUTCOMES:
Listening Effort as assessed by the Adaptive Categorical Listening Effort Scaling (ACALES) | Data is collected during the second lab visit for each participant, approximately 2 weeks after study enrollment. The duration of the study visit including testing is approximately 2.5 hours.
  The ACALES is an adaptive measure of listening effort where the target and interfering background signals are adapted according to participant feedback. Following the target presentation, participants rate listening effort on a 14-point scale

OTHER OUTCOMES:
Hearing Instrument Device Preference Questionnaire | Data is collected during the second lab visit for each participant, approximately 2 weeks after study enrollment. The duration of the study visit including testing is approximately 2.5 hours.
  Participants are asked to subjectively rate elements of sound quality and overall preference of the devices under test following standardized presentation of speech-in-noise stimuli in the lab environment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida Auditory Neurosciences & Technology Lab, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No